CLINICAL TRIAL: NCT05490004
Title: Evaluating an Educational Intervention for Improving Provider Recognition and Response to Intimate Partner Violence (IPV) Experienced by Veterans and Their Families - A Mixed Method Pilot Randomized Trial
Brief Title: RISE With Veteran Service Providers
Acronym: RISE Vet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Atlas Institute for Veterans and Families (Unknown)
Responsible Party: Principal Investigator, Melissa Kimber, PhD, MSW, RSW, Assistant Professor, Department of Psychiatry & Behavioural Neurosciences, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HiREB # 14243
Record Dates: First submitted 2022-07-28; First posted 2022-08-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Domestic Violence; Veterans Family; Veterans; Child Maltreatment
Keywords: Family Violence; Medical Education; Education Scholarship; Health Professions Education; Mandatory Reporting; Child Maltreatment; Intimate Partner Violence; Veterans; Veterans Family
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Intervention Model Description: To determine the feasibility of evaluating the effectiveness of both of VEGA's educational approaches, as well as to generate preliminary estimates of effect for sampling and effect size calculations, a two-arm pilot randomized controlled trial (RCT) will be used (Eldridge et al., 2016). Eligible participants will be randomly assigned to receive either self-directed (i.e., experimental) or facilitator-led (i.e., active control (AC)) VEGA.
Who Masked: Outcomes Assessor
Masking Description: The Research Assistant will be blinded to group allocation. The RA will be responsible for following-up with participants to make sure they've completed quantitative assessments (online survey) or, if participants choose to complete the surveys over the phone, the RA will complete them over the phone with the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Facilitator-Led VEGA (Active Comparator): Facilitator-led VEGA uses a group-based approach where participants complete the Violence, Evidence, Guidance, Action Project (VEGA) content as a virtual or face-to-face workshop (i.e., facilitator-led VEGA). In this study, all workshops will be virtual to prevent social gathering during COVID-19.
  If a participant is randomized to this arm, the active control arm, they will be informed that they need to attend a facilitator-led VEGA session via virtual workshop format. The AC intervention will be facilitated via Zoom technology, by two trained facilitators with between 10 to 20 participants in each workshop (keeping the recommended 10:1 participant-to-facilitator ratio) and will last approximately 3 hours. The workshop approach is delivered by trained facilitators and is standardized via the use of a flexibly structured facilitator's guide. Facilitator-led VEGA will deliver material didactically with synchronous lecturing, use case-based role play, and include group-based polling.
  Interventions: Other: Violence, Evidence, Guidance, Action Project (VEGA) Education Intervention
- Self-Directed VEGA (Experimental): Self-directed VEGA uses an approach where participants complete the Violence, Evidence, Guidance, Action Project (VEGA) content online as a self-directed educational activity, at their own pace in a series of modules. Individuals will register to access the VEGA Education Resources site. Participants have the option of completing the self-directed VEGA arm in either English or French as the VEGA Educational Resources site offers the content in French and English.
  If a participant is randomized to the experimental arm, they will be asked to complete the self-directed VEGA at their convenience, within one week of when they are informed they have been asked to complete the self-directed VEGA program. It will take approximately 3 hours for participants to complete all modules.
  Participants will read didactic material, complete case-based animated simulations, and complete individual multiple-choice questions with response feedback.
  Interventions: Other: Violence, Evidence, Guidance, Action Project (VEGA) Education Intervention

INTERVENTIONS:
Other: Violence, Evidence, Guidance, Action Project (VEGA) Education Intervention — VEGA is a novel education intervention that has the potential to improve the preparation of healthcare and social service providers (HHSPs) to be able to effectively recognize and respond to intimate partner violence (IPV) and related forms of family violence, including child maltreatment (CM), in their clinical encounters. VEGA was developed based on systematic reviews and consultation with individuals belonging to 22 national healthcare and social service organizations, including the Royal College of Physicians and Surgeons of Canada. VEGA follows a competency-based framework and a participatory, encounter-based curriculum that includes four learning modules: (a) the epidemiology of IPV and CM; (b) strategies for safely recognizing and responding to (i) IPV and (ii) CM; and (c) principles for ensuring safe clinical encounters for IPV and CM discussions.
  Other Names: VEGA Family Violence Education Resources

SUMMARY:
Veterans and their families are more likely to experience forms of family violence like intimate-partner violence and child maltreatment. Evidence suggests that healthcare and social service providers (HSSPs) need more training to effectively and confidently recognize and respond to these situations. The Violence, Evidence, Guidance, Action (VEGA) Educational Intervention is a novel education intervention aimed at improving provider's preparation for these clinical encounters. The goal of this project is to determine the acceptability and feasibility of a future randomized-controlled trial comparing two approaches (facilitator-led VEGA or self-directed VEGA) to administering the VEGA training to understand whether/how these approaches can support HSSPs continued care of veterans and their families. The investigators aim to generate initial estimates of the effectiveness of both approaches in improving HSSPs knowledge and skills to effectively recognize and respond to intimate-partner violence and related forms of family violence, including child maltreatment. As well, the investigators aim to contribute to the knowledge base regarding optimal educational approaches for HSSP education in family violence.

The investigators hypothesize that there will be significant increases in preparedness, knowledge and skills, and self-efficacy to recognize and respond to both CM and IPV in both the experimental and AC arms from Time 1 (baseline) to Time 2 (immediately after the intervention) and Time 1 (baseline) to Time 3 (3 month follow-up). These improvements will be slightly attenuated in the experimental arm. Qualitative data pertaining to perceived value and impact will corroborate the quantitative findings.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a regulated healthcare or social service provider that is an active member in good standing with the associated regulatory college.
* Participant is fluent in written and spoken English.
* We are looking for participants who are currently working with or have previous experience working with military and/or RCMP veterans or their family members. Participants must meet one of the following criteria:

  1. Participant works with military and/or RCMP veterans or family members of military and/or RCMP veterans in a direct service capacity at least one day per week OR
  2. Participant has two years or more of experience working with military and/or RCMP veterans or family members of military and/or RCMP veterans in a direct service capacity OR
  3. Participant has worked with 15 or more patients that were either military and/or RCMP veterans or family members of military and/or RCMP veterans in a direct service capacity.

Exclusion Criteria:

* Participant has previously accessed VEGA intervention materials.
* Participant is currently enrolled in or plans to enroll in any other educational intervention focused on family violence within the study time period (approximately next 3 months).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Number of Providers Who Meet Eligibility Criteria | Through study completion, an average of 4 months
  The RC will track the number of providers who meet eligibility criteria, our aims are that we will recruit a total of 80 participants within 16 weeks, an average of 5 providers per week.
Number of Providers who Consent | Through study completion, an average of 4 months
  The RC will track the number of providers who consent to the study and agree to be randomized to either self-directed or facilitator-led VEGA education approaches, both overall and per week of recruitment. Our aim is that the proportion of providers who contact the research team about participation and who consent to randomization will be 70% or greater.
Number of Providers who Complete Assigned Intervention | Through study completion, an average of 4 months
  The RC will track the proportion of providers who are randomized and complete each arm, with completion consisting of reviewing all module content and the animated simulations in the case of self-directed VEGA and full attendance of the virtual workshop in the case of facilitator-led VEGA. Our goal is that the proportion of providers who are randomized and complete the assigned intervention will be 70% or greater for each arm. The acceptability of the facilitator-led and self-directed educational approaches as well as their value and impact will be determined via the coding of qualitative interview data from a sub-sample of participants.
Number of Providers who Complete Assessments | Through study completion, an average of 4 months
  The RC will track the feasibility of collecting trial outcome data (survey assessments) at Time 1, Time 2, and Time 3. Our goal is that the proportion of missing data for each time point will be less than 20%. Qualitative description will be used to expand and extend what we learn about acceptability and feasibility of implementing the associated research activities, we anticipate participants will not identify any fatal flaws related to the conduct of an RCT.

SECONDARY OUTCOMES:
Child Maltreatment Vignette Scale | Time 1 (one week before intervention), Time 2 (immediately after the intervention), Time 3 (3 month follow-up)
  Child Maltreatment Vignette scale (Pelletier et al., 2014; Pelletier & Knox, 2017) is a psychometrically validated measure of knowledge and skill accuracy related to recognizing and responding to child maltreatment. Respondents will be prompted to review 14 distinct analog vignettes that depict a range of signs and symptoms of possible CM exposure and asked if they suspect child maltreatment and if they would report to Child Welfare Services. Changes to the question wording and small changes to the wording of the scenarios were made to align the measure with the Canadian context. A mean "knowledge and skill accuracy" score will be produced for analysis, with higher scores indicative of greater knowledge and skill accuracy related to CM. In a future RCT, this would be one of the primary outcomes of interest since this is a robust measure of practitioner knowledge and skills related to CM.
Child Maltreatment Knowledge and Skills Questions (Developed by VEGA Team) | Time 1 (one week before intervention), Time 2 (immediately after the intervention), Time 3 (3 month follow-up)
  Participants will be asked a series of questions about their knowledge and skills related to recognizing and responding to child maltreatment. These were developed by the VEGA training research team to capture specific aspects of child maltreatment knowledge directly addressed in the VEGA intervention and which are outside the scope of the child maltreatment vignette scale. The questions ask about the following topics (and more not mentioned here): parental/family risk factors for family violence, what future outcomes are associated with child maltreatment, other possible signs of child abuse, and principles for good documentation and providing ongoing care to children experiencing maltreatment. Including this measure in our study will allow us to make cross sample comparisons.
The Physician Readiness to Manage Intimate Partner Violence Survey: IPV Knowledge | Time 1 (one week before intervention), Time 2 (immediately after the intervention), Time 3 (3 month follow-up)
  The Physician Readiness to Manage Intimate Partner Violence Survey (PREMIS) is a 67-item self-report tool that was developed to assess physician management of intimate partner violence across 10 subscales (Short et al., 2006; Connor et al., 2011). The IPV knowledge section, consisting of multiple answer, multiple choice, and true-false questions will be used to measure IPV knowledge and skills. An IPV "knowledge score" will be computed following previous scoring guidelines (Short et al., 2006). In a future RCT, this would be a primary outcome of interest to measure practitioner knowledge and skills related to IPV.
The Physician Readiness to Manage Intimate Partner Violence Survey: Preparedness Subscale | Time 1 (one week before intervention), Time 2 (immediately after the intervention), Time 3 (3 month follow-up)
  The preparedness subscale of PREMIS asks respondents to indicate the extent to which they feel prepared to address various aspects of IPV recognition and response when working with their clients across 10 items; these aspects include the conduct of safety assessments, asking appropriate questions about IPV, responding to IPV disclosures, among others. Response options are on a 7-item Likert type scale ranging from "Not prepared" (1) to "Quite Well Prepared" (7) and items are averaged to generate a mean score for practitioner preparedness, with higher scores indicative of generally greater preparedness to recognize and respond to IPV. For the purposes of this study, two adapted versions of the preparedness subscale were used to assess preparedness to recognize and respond to IPV and CM.
The Physician Readiness to Manage Intimate Partner Violence Survey: Opinions | Time 1 (one week before intervention), Time 3 (3 month follow-up)
  The Opinions section of the PREMIS asks respondents to indicate their level of agreement/disagreement with various statements about care of those with IPV across 32 items. Response options are on a 7-item Likert type scale ranging from (1) Strongly Disagree to (7) Strongly Agree. Our adapted version will be used to measure provider attitudes and beliefs about IPV and care of those with IPV in five subscales: (1) preparation, (2) workplace issues, (3) self-efficacy (which will also be assessed at Time 2), (4) alcohol/drugs, and (5) victim understanding. We will follow previous methods to calculate these subscales by averaging the responses to items that make up the subscale (Short et al., 2006). The three items comprising the self-efficacy subscale will be a primary outcome of interest in a future RCT as a measure of provider's self-efficacy to recognize and respond to IPV.
Mandatory Reporting Self-Efficacy Scale (MRSES) | Time 1 (one week before intervention), Time 2 (immediately after the intervention), Time 3 (3 month follow-up)
  The MRSES is a 7-item self-report measure that asks respondents to indicate the extent to which they perceive their ability to implement a series of behaviours related to mandatory reporting of CM (Ayling, 2019). Informed by Bandura's self-efficacy theory and recommendations for self-efficacy scales (Bandura, 2006), response options are anchored on a scale from 0 to 100 with: "cannot do at all (0)"; moderately can do (50)"; and "highly certain can do (100)." A total score is generated by summing items across the scale for each participant, with higher scores indicative of greater self-efficacy related to recognizing and reporting suspected CM. We anticipate that this measure will be a key mediator of interest in a future definitive RCT given that across provincial and territorial jurisdictions in Canada (including Ontario), a suspicion of CM meets the threshold for a report to child protection authorities (Dubowitz, 2014; Mathews and Kenny, 2008).
Brief Individual Readiness for Change Scale | Time 1 (one week before intervention), Time 2 (immediately after the intervention)
  The Brief Individual Readiness for Change (BIRCS) scale is a 5-item readiness for change tool (Goldman, 2009). The scale's purpose is to screen for practitioners' readiness for change, in other words their receptivity to learning and applying new evidence-based research practices. For the purpose of this study, the items were adapted to assess provider's readiness to recognize and respond to all forms of (a) IPV and (b) CM in their practice. Response options range from '0' Strongly Disagree to '4' Strongly Agree. Two items were added, "I believe recognizing and responding to [IPV/CM] in my practice improves outcomes for my clients," and "I am motivated to learn about [IPV/CM]" to capture other aspects of providers' readiness to learn about IPV and CM and their belief's about how this will impact their practice.

OTHER OUTCOMES:
Previous Training in Intimate Partner Violence and Child Maltreatment | Time 1 (one week before intervention)
  Participants will be asked questions to gauge their previous education or training in IPV and CM. Participants will be given a definition of IPV and CM and asked in what subject areas of IPV and CM they have received education and training in, and which of these environments (up to three) have been the most helpful.
Thoughts and Beliefs about Recognizing and Responding to IPV and CM in Professional Roles | Time 1 (one week before intervention), Time 2 (immediately after the intervention)
  Participants will be asked to rate their agreement with four statements asking how much they believe (1) recognizing IPV (2) recognizing CM (3) responding to IPV and (4) responding to CM is a part of their professional role. We will report, on average across the sample, how participants rate their agreement on a Likert scale for statements 1-4. We are recruiting a wide variety of HHSPs that we anticipate may vary in their self-perceptions of how relevant recognizing and responding to IPV and CM is in their professional roles. In qualitative interviews we will ask participants how often they believe they will encounter family violence in their practice (and how relevant it is to their professional role), the purpose of this outcome measure is to gauge this in our entire sample.
Satisfaction with VEGA Training | Time 2 (immediately after the intervention)
  Participants will complete a series of multiple choice and short-answer questions asking what they thought about the VEGA training. These questions will apply to all participants whether they completed self-directed or facilitator-led VEGA. Questions will include whether they believe the intended learning outcomes were achieved, what they thought of the instructional materials and educational scenarios, and how they would rate the usefulness of VEGA.
Demographics | Pre-Intervention
  Sociodemographic characteristics will be collected for all participants who are screened for the study, whether they are ineligible or eligible. These will include their age, province of practice, highest level of education attainment, their major discipline, their sex at birth and their self-identified gender. We will also collect some characteristics about the current organization they work for, specifically what populations among military and/or RCMP veterans and their families they serve and if consent is required by the veteran for the participant to provide services to a family member.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Kimber, PhD, MSW, RSW, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Requests for data for analyses (e.g. by Research Team Members, graduate trainees) will be managed by the research coordinator and overseen by the PI, including Dr. Melissa Kimber. This will not include identifying information of participants, only de-identified data would be shared.

REFERENCES:
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Pelletier HL, Knox M. Incorporating Child Maltreatment Training into Medical School Curricula. J Child Adolesc Trauma. 2017;10(3):267-274. doi: 10.1007/s40653-016-0096-x. Epub 2016 May 12. PMID 29026450
- [Background] Connor PD, Nouer SS, Mackey ST, Tipton NG, Lloyd AK. Psychometric properties of an intimate partner violence tool for health care students. J Interpers Violence. 2011 Mar;26(5):1012-35. doi: 10.1177/0886260510365872. Epub 2010 Jun 28. PMID 20587479
- [Background] Short LM, Alpert E, Harris JM Jr, Surprenant ZJ. A tool for measuring physician readiness to manage intimate partner violence. Am J Prev Med. 2006 Feb;30(2):173-180. doi: 10.1016/j.amepre.2005.10.009. PMID 16459217
- [Background] Mathews B, Kenny MC. Mandatory reporting legislation in the United States, Canada, and Australia: a cross-jurisdictional review of key features, differences, and issues. Child Maltreat. 2008 Feb;13(1):50-63. doi: 10.1177/1077559507310613. PMID 18174348
- [Background] Afifi TO, Taillieu T, Zamorski MA, Turner S, Cheung K, Sareen J. Association of Child Abuse Exposure With Suicidal Ideation, Suicide Plans, and Suicide Attempts in Military Personnel and the General Population in Canada. JAMA Psychiatry. 2016 Mar;73(3):229-38. doi: 10.1001/jamapsychiatry.2015.2732. PMID 26817953
- [Background] Afifi TO, Sareen J, Taillieu T, Stewart-Tufescu A, Mota N, Bolton SL, Asmundson GJG, Enns MW, Ports KA, Jetly R. Association of Child Maltreatment and Deployment-related Traumatic Experiences with Mental Disorders in Active Duty Service Members and Veterans of the Canadian Armed Forces: Association de la Maltraitance des Enfants et des Experiences Traumatisantes Liees au Deploiement Avec les Troubles Mentaux Chez les Membres du Service Actif et Les Anciens Combattants des Forces Armees Canadiennes. Can J Psychiatry. 2021 Nov;66(11):961-970. doi: 10.1177/0706743720987086. Epub 2021 Jan 21. PMID 33472392
- [Background] Marshall AD, Panuzio J, Taft CT. Intimate partner violence among military veterans and active duty servicemen. Clin Psychol Rev. 2005 Nov;25(7):862-76. doi: 10.1016/j.cpr.2005.05.009. PMID 16006025
- [Background] Sparrow K, Kwan J, Howard L, Fear N, MacManus D. Systematic review of mental health disorders and intimate partner violence victimisation among military populations. Soc Psychiatry Psychiatr Epidemiol. 2017 Sep;52(9):1059-1080. doi: 10.1007/s00127-017-1423-8. Epub 2017 Jul 26. PMID 28748307
- [Background] Griffith J, J Bryan C. Deployment Experiences and Suicidal Behaviors Related to Interpersonal Violence Perpetration Among Army National Guard Soldiers. Violence Vict. 2020 Dec 1;35(6):841-860. doi: 10.1891/VV-D-18-00174. PMID 33372113
- [Background] Zamorski MA, Wiens-Kinkaid ME. Cross-sectional prevalence survey of intimate partner violence perpetration and victimization in Canadian military personnel. BMC Public Health. 2013 Oct 28;13:1019. doi: 10.1186/1471-2458-13-1019. PMID 24165440
- [Background] MacMillan HL, Kimber M, Stewart DE. Intimate Partner Violence: Recognizing and Responding Safely. JAMA. 2020 Sep 22;324(12):1201-1202. doi: 10.1001/jama.2020.11322. No abstract available. PMID 32960228
- [Background] Stewart DE, MacMillan H, Kimber M. Recognizing and Responding to Intimate Partner Violence: An Update. Can J Psychiatry. 2021 Jan;66(1):71-106. doi: 10.1177/0706743720939676. Epub 2020 Aug 10. No abstract available. PMID 32777936
- [Background] Beynon CE, Gutmanis IA, Tutty LM, Wathen CN, MacMillan HL. Why physicians and nurses ask (or don't) about partner violence: a qualitative analysis. BMC Public Health. 2012 Jun 21;12:473. doi: 10.1186/1471-2458-12-473. PMID 22721371
- [Background] Kimber M, McTavish JR, Couturier J, Le Grange D, Lock J, MacMillan HL. Identifying and responding to child maltreatment when delivering family-based treatment-A qualitative study. Int J Eat Disord. 2019 Mar;52(3):292-298. doi: 10.1002/eat.23036. Epub 2019 Feb 6. PMID 30729594
- [Background] Kimber M, McTavish JR, Luo C, Couturier J, Dimitropoulos G, MacMillan H. Mandatory reporting of child maltreatment when delivering family-based treatment for eating disorders: A framework analysis of practitioner experiences. Child Abuse Negl. 2019 Feb;88:118-128. doi: 10.1016/j.chiabu.2018.11.010. Epub 2018 Nov 23. PMID 30476720
- [Background] McTavish JR, Kimber M, Devries K, Colombini M, MacGregor JCD, Wathen CN, Agarwal A, MacMillan HL. Mandated reporters' experiences with reporting child maltreatment: a meta-synthesis of qualitative studies. BMJ Open. 2017 Oct 16;7(10):e013942. doi: 10.1136/bmjopen-2016-013942. PMID 29042370
- [Background] Alnasser Y, Albijadi A, Abdullah W, Aldabeeb D, Alomair A, Alsaddiqi S, Alsalloum Y. Child maltreatment between knowledge, attitude and beliefs among Saudi pediatricians, pediatric residency trainees and medical students. Ann Med Surg (Lond). 2017 Feb 21;16:7-13. doi: 10.1016/j.amsu.2017.02.008. eCollection 2017 Apr. PMID 28275426
- [Background] Inanici SY, Celik E, Hidiroglu S, Ozdemir M, Inanici MA. Factors associated with physicians' assessment and management of child abuse and neglect: A mixed method study. J Forensic Leg Med. 2020 Jul;73:101972. doi: 10.1016/j.jflm.2020.101972. Epub 2020 May 30. PMID 32658746
- [Background] Flaherty EG, Sege R, Price LL, Christoffel KK, Norton DP, O'Connor KG. Pediatrician characteristics associated with child abuse identification and reporting: results from a national survey of pediatricians. Child Maltreat. 2006 Nov;11(4):361-9. doi: 10.1177/1077559506292287. PMID 17043321
- [Background] Flaherty EG, Sege R, Binns HJ, Mattson CL, Christoffel KK. Health care providers' experience reporting child abuse in the primary care setting. Pediatric Practice Research Group. Arch Pediatr Adolesc Med. 2000 May;154(5):489-93. doi: 10.1001/archpedi.154.5.489. PMID 10807301
- [Background] Regnaut O, Jeu-Steenhouwer M, Manaouil C, Gignon M. Risk factors for child abuse: levels of knowledge and difficulties in family medicine. A mixed method study. BMC Res Notes. 2015 Oct 30;8:620. doi: 10.1186/s13104-015-1607-9. PMID 26514128
- [Background] Flaherty EG, Sege R. Barriers to physician identification and reporting of child abuse. Pediatr Ann. 2005 May;34(5):349-56. doi: 10.3928/0090-4481-20050501-08. PMID 15948346
- [Background] Norman GR, Sloan JA, Wyrwich KW. The truly remarkable universality of half a standard deviation: confirmation through another look. Expert Rev Pharmacoecon Outcomes Res. 2004 Oct;4(5):581-5. doi: 10.1586/14737167.4.5.581. PMID 19807551
- [Background] Crowe M, Inder M, Porter R. Conducting qualitative research in mental health: Thematic and content analyses. Aust N Z J Psychiatry. 2015 Jul;49(7):616-23. doi: 10.1177/0004867415582053. Epub 2015 Apr 21. PMID 25900973
- [Background] Guetterman TC, Fetters MD, Creswell JW. Integrating Quantitative and Qualitative Results in Health Science Mixed Methods Research Through Joint Displays. Ann Fam Med. 2015 Nov;13(6):554-61. doi: 10.1370/afm.1865. PMID 26553895
- [Background] Flaherty EG, Sege R, Mattson CL, Binns HJ. Assessment of suspicion of abuse in the primary care setting. Ambul Pediatr. 2002 Mar-Apr;2(2):120-6. doi: 10.1367/1539-4409(2002)0022.0.co;2. PMID 11926843
- [Background] Vaismoradi M, Turunen H, Bondas T. Content analysis and thematic analysis: Implications for conducting a qualitative descriptive study. Nurs Health Sci. 2013 Sep;15(3):398-405. doi: 10.1111/nhs.12048. Epub 2013 Mar 11. PMID 23480423
- [Derived] Kimber M, Baker-Sullivan E, Stewart DE, Vanstone M. Improving Health Professional Recognition and Response to Child Maltreatment and Intimate Partner Violence: Protocol for Two Mixed Methods Pilot Randomized Controlled Trials. JMIR Res Protoc. 2024 Mar 21;13:e50864. doi: 10.2196/50864. PMID 38512307
- See also: This is the VEGA Project website, where the public can access VEGA Family Violence Education Resources. More information can be found here about the development of VEGA. — https://vegaproject.mcmaster.ca/